CLINICAL TRIAL: NCT04767828
Title: A Single Arm Study of Brain Metastasis in Patients With HER2-positive Breast Cancer Treated With Pyrrolidine Maleate and Capecitabine Combined With Brain Radiotherapy
Brief Title: A Single Arm Study of Brain Metastasis in Patients With HER2-positive Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2019316
Record Dates: First submitted 2021-02-05; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: TTP
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One arm exploratory research (Experimental): Brain radiation therapy: the dose and frequency of brain radiation therapy are determined by the doctor according to the patient's condition. Pyrrotini: 400 mg once a day, oral within 30 minutes after breakfast for 21 days. Cassitabine: twice a day, 800 mg / m2 orally within 30 minutes after each meal (one morning and one night, 12 hours apart, equivalent to a daily dose of 1600 mg / m2, one dose in the morning and one dose in the morning)
  Interventions: Drug: PYRROTINI; Radiation: Brain radiation therapy

INTERVENTIONS:
Drug: PYRROTINI — CAPECITABINE: 800 mg/m2 twice daily, taken orally within 30 minutes after meal (one in the morning and one in the evening, 12 hours apart, equal to a daily dose of 1600 mg/m2, with one dose in the morning and one dose in the morning) .
  Other Names: CAPECITABINE
Radiation: Brain radiation therapy — Brain radiation therapy: the dose and frequency of brain radiation therapy are determined by the doctor according to the patient's condition.

SUMMARY:
The aim of this study was to evaluate the progression time and efficacy of brain tumors in patients with brain metastases from HER2-positive breast cancer treated with Pyrrolidine and Capecitabine combined with brain radiotherapy.

DETAILED DESCRIPTION:
Brain metastases are very common in HER2-positive breast cancer patients. The vast majority of patients with metastatic brain tumors are in advanced stages of the disease. If not treated in time, the natural course of the disease is extremely short. At present, the main treatment of brain metastases from breast cancer is radiotherapy, combined with chemotherapy and targeted therapy drugs. On the basis of previous clinical studies, the aim of this study was to explore the efficacy and safety of combined brachytherapy with Pyrrotidine and Capecitabine in patients with brain metastases from HER2-positive breast cancer, in order to provide a new, safer and more effective treatment for patients with brain metastases from breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to enrollment.
2. Age 18-75 years, female.
3. Patients with pathologically confirmed HER2 expression-positive breast cancer brain metastases; HER2 expression-positive refers to those with a standard immunohistochemical staining (IHC) test showing HER2 as 3+ and/or fluorescence in situ hybridization technique (FISH) positive (confirmed by investigator review at their trial center).
4. The presence of CNS lesions as confirmed by cranial CT or MRI.
5. ECOG score: 0 to 2.
6. Expected survival of not less than 12 weeks.
7. having received no previous brain radiotherapy or having received brain radiotherapy at the dose specified in the trial protocol.
8. Patients who have been on pyrrolizidine for ≤ 3 months after diagnosis of brain metastases and whose disease has not progressed.
9. The function of vital organs meets the following requirements (excluding the use of any blood components and cell growth factors within 14 days).

   A) Routine blood examination criteria need to be met: Hb ≥ 100 g/L; ANC ≥ 1.5×109 /L; PLT ≥ 75×109 /L B) Biochemical examination should meet the following criteria: TBIL≤1.5×ULN (upper limit of normal); ALT and AST≤2.5×ULN; ALT and AST≤5×ULN if liver metastasis; serum creatinine≤1.5×ULN, creatinine clearance≥50ml/min (based on Cockroft and Gault formula) C) Cardiac ultrasound; left ventricular ejection fraction (LVEF) ≥ 50%
10. Female patients who are non-surgically sterilized or of childbearing age are required to use a medically approved form of contraception (e.g., IUD, pill, or condom) during and for 3 months after the end of the study treatment period; female patients of childbearing age who are non-surgically sterilized must have a negative serum or urine HCG test within 7 days prior to study enrollment; and must be non-lactating.
11. Subjects are voluntarily enrolled in the study, are compliant, and cooperate with safety and survival follow-up.

Exclusion Criteria:

1. Presence of third interstitial fluid that cannot be controlled by drainage or other methods, such as massive pleural and ascites fluid.
2. the presence of multiple factors that interfere with oral administration and absorption of the drug (e.g., inability to swallow, post-gastrectomy, chronic diarrhea, and intestinal obstruction).
3. have a proven allergy to the drug components of this regimen.
4. Patients who are known to be pregnant or planning to become pregnant, or patients of gestational age who are unwilling to use effective contraception throughout the trial period.
5. Patients with severe concomitant disease or who, in the opinion of the investigator, are not suitable for inclusion.
6. Patients with the presence of meningeal metastases.
7. having participated in a clinical trial of another drug within 4 weeks prior to enrollment.
8. Patients who have used capecitabine during the neoadjuvant/adjuvant phase of therapy are allowed to be enrolled, but those who are ineffective or cannot tolerate capecitabine during the neoadjuvant/adjuvant phase of therapy need to be excluded; patients who have used capecitabine for ≤ 3 months after brain metastasis and whose disease has not progressed can be enrolled; other drugs for which the active ingredient is 5-fluorouracil are treated as capecitabine (Note: " used capecitabine" refers to continuous standardized use of capecitabine for ≥ 2 cycles).
9. Concurrently receiving other antitumor therapy.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 43 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Time of intracranial tumor progression | through study completion, an average of 1 year
  Objective to evaluate the intracranial tumor progression time of piratinib and capecitabine combined with brain radiotherapy for HER2 positive breast cancer patients with brain metastasis

SECONDARY OUTCOMES:
Progression-free survival | through study completion, an average of 1 year
  Objective to evaluate the progression free survival (PFS) of pirotinib and capecitabine combined with brain radiotherapy in HER2 positive breast cancer patients with brain metastasis.
Objective remission rate | through study completion, an average of 1 year
  objective response rate (ORR) of pirotinib and capecitabine combined with brain radiotherapy in HER2 positive breast cancer patients with brain metastasis.
Duration of treatment effect | throughout studythrough study completion, an average of 1 year
  Duration of treatment effect (DCR) of pirotinib and capecitabine It refers to the time between the first assessment of CR or PR and the first assessment of PD (Progressive Disease) or death from any causecombined with brain radiotherapy in HER2 positive breast cancer patients with brain metastasis.
Disease control rate | throughout studythrough study completion, an average of 1 year
  Objective to evaluate the disease control rate of pirotinib and capecitabine combined with brain radiotherapy in HER2 positive breast cancer patients with brain metastasis
Clinical Benefit Rate | throughout studythrough study completion, an average of 1 year
  Objective to evaluate the clinical benefit rate of pirotinib and capecitabine combined with brain radiotherapy in HER2 positive breast cancer patients with brain metastasis
Overall survival | through study completion, an average of 1 year
  Objective to evaluate the overall survival of piratinib and capecitabine combined with brain radiotherapy in HER2 positive breast cancer patients with brain metastasis
Graded healing assessment | through study completion, an average of 1 year
  Objective to evaluate the effect of pyrrolotinib and capecitabine combined with brain radiotherapy in patients with HER2 positive breast cancer with brain metastasis，The score of graded healing assessment was 0-4. The higher the score, the better the result

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, MD, Principal Investigator — 研究者
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China